CLINICAL TRIAL: NCT05333757
Title: Assessing the Quality of Life in Adults With Spinal Deformity: a Retrospective Comparison Between Two Questionnaires
Brief Title: Assessing the Quality of Life in Adults With Spinal Deformity
Status: Completed | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: A-ISYQOL
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Scoliosis; Quality of Life
MeSH Terms: conditions — Scoliosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of life: Adult patients treated conservatively for idiopathic scoliosis or undergoing clinical monitoring who have completed both questionnaires at least once and simultaneously and who meet the following inclusion criteria:
  * Age ≥ 18 years
  * Diagnosis of idiopathic or degenerative scoliosis with curve ≥30 ° Cobb
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Adults with spinal deformities were asked to complete two questionnaires assessing quality of life

SUMMARY:
Spinal deformities, such as scoliosis, can have a significant impact on the physical and psychological health of patients. Over time, specific tools for this condition have been developed to investigate the extent of this impact, such as the SRS-22 questionnaire and ISYQOL questionnaire.

The latter was initially used for underage patients, but given that some of them continue their therapy and the monitoring beyond the age of 18, we have continued its use in these subjects as well. Given the clinical usefulness and given the lack of questionnaires developed in the Rasch environment for adults, we have extended the application of the ISYQOL questionnaire to the adult population. However, a comparison between the ISYQOL and SRS-22 in adults has not yet been made.

The objective of this study is to verify the validity of ISYQOL and to compare the properties of ISYQOL with those of the SRS-22 questionnaire in adults with spinal deformity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of idiopathic or degenerative scoliosis with ≥30 ° Cobb curve

Exclusion Criteria:

* Previous spinal surgery
* Previous and relevant illnesses, surgery or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated conservatively for idiopathic scoliosis or undergoing clinical monitoring
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Statistical properties of SRS-22 and ISYQOL questionnaire | through study completion, an average of 1 year
  The Spearman correlation coefficient will be used to evaluate the concurrent validity of ISYQOL questionnaire. Cronbach's alpha will be used to evaluate the internal validity of ISYQOL questionnaire.
  Rasch analysis will be applied to explore the characteristics of the two tools. In addition, the reproducibility of the measurement. Usually, the goal is to obtain a reliability> 0.8.

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be uploaded to public repository